CLINICAL TRIAL: NCT07307807
Title: Evaluation of Postoperative Pain and Lesion Healing in Periapical Lesion-Affected Teeth Obturated With Different Root Canal Sealers: Prospective Study
Brief Title: Evaluation of Postoperative Pain and Lesion Healing in Periapical Lesion-Affected Teeth Obturated With Different Root Canal Sealers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Neslihan Büşra Keskin, Assoc. Prof., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/14-03(KA-25010)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Root Canal Obturation; Apical Periodontitis
Keywords: AH Plus; TotalFill BC Sealer; Postoperative pain; Fractal analysis; Visual Analog Scale (VAS)
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The bioistatician performing the data analysis will be blinded to group allocation. The clinician performing the treatments will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AH Plus and PAI 2-3 (Experimental): Teeth with PAI scores of 2 and 3 that were obturated with AH Plus and completed in a single visit.
  Interventions: Procedure: AH Plus and PAI 2-3
- AH Plus and PAI 4 (Experimental): Teeth with a PAI score of 4 that were obturated with AH Plus and completed in a single visit.
  Interventions: Procedure: AH Plus and PAI 4
- TotalFill BC Sealer and PAI 2-3 (Experimental): Teeth with PAI scores of 2 and 3 obturated with TotalFill BC and completed in a single visit.
  Interventions: Procedure: TotalFill BC Sealer and PAI 2-3
- TotalFill BC Sealer and PAI 4 (Experimental): Teeth with a PAI score of 4 obturated with TotalFill BC and completed in a single visit.
  Interventions: Procedure: TotalFill BC Sealer and PAI 4

INTERVENTIONS:
Procedure: AH Plus and PAI 2-3 — The AH Plus root canal sealer, mixed in accordance with the manufacturer's instructions, will be applied together with master cones into root canals with PAI scores of 2-3. Control periapical radiographs will be obtained to evaluate the quality of the root canal fillings.
  Volunteers will be asked to record the pain they experience before treatment and at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as 1 week after treatment, using a Visual Analog Scale (VAS) form. One week after treatment, volunteers will be contacted by telephone, and the pain scores recorded on the pain assessment forms will be entered into the patient records. Six months after completion of the endodontic treatment, volunteers will be contacted by telephone and recalled for follow-up. Control periapical radiographs will be obtained from the volunteers, and healing will be evaluated.
  Arms: AH Plus and PAI 2-3
Procedure: AH Plus and PAI 4 — The AH Plus root canal sealer, mixed in accordance with the manufacturer's instructions, will be applied together with master cones into root canals with PAI score of 4. Control periapical radiographs will be obtained to evaluate the quality of the root canal fillings.
  Volunteers will be asked to record the pain they experience before treatment and at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as 1 week after treatment, using a Visual Analog Scale (VAS) form. One week after treatment, volunteers will be contacted by telephone, and the pain scores recorded on the pain assessment forms will be entered into the patient records.
  Six months after completion of the endodontic treatment, volunteers will be contacted by telephone and recalled for follow-up. Control periapical radiographs will be obtained from the volunteers, and healing will be evaluated
  Arms: AH Plus and PAI 4
Procedure: TotalFill BC Sealer and PAI 2-3 — The TotalFill BC root canal sealer, mixed in accordance with the manufacturer's instructions, will be applied together with master cones into root canals with PAI scores of 2-3. Control periapical radiographs will be obtained to evaluate the quality of the root canal fillings.
  Volunteers will be asked to record the pain they experience before treatment and at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as 1 week after treatment, using a Visual Analog Scale (VAS) form. One week after treatment, volunteers will be contacted by telephone, and the pain scores recorded on the pain assessment forms will be entered into the patient records.
  Six months after completion of the endodontic treatment, volunteers will be contacted by telephone and recalled for follow-up. Control periapical radiographs will be obtained from the volunteers, and healing will be evaluated.
  Arms: TotalFill BC Sealer and PAI 2-3
Procedure: TotalFill BC Sealer and PAI 4 — The AH Plus root canal sealer, mixed in accordance with the manufacturer's instructions, will be applied together with master cones into root canals with PAI score of 4. Control periapical radiographs will be obtained to evaluate the quality of the root canal fillings.
  Volunteers will be asked to record the pain they experience before treatment and at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as 1 week after treatment, using a Visual Analog Scale (VAS) form. One week after treatment, volunteers will be contacted by telephone, and the pain scores recorded on the pain assessment forms will be entered into the patient records.
  Six months after completion of the endodontic treatment, volunteers will be contacted by telephone and recalled for follow-up. Control periapical radiographs will be obtained from the volunteers, and healing will be evaluated.
  Arms: TotalFill BC Sealer and PAI 4

SUMMARY:
The root canal treatment of volunteers with asymptomatic apical periodontitis will be completed using TotalFill BC and AH Plus root canal sealers, and postoperative pain as well as healing will be comparatively evaluated through radiographic follow-ups at predetermined time intervals.

DETAILED DESCRIPTION:
The study is planned as a randomized controlled clinical trial. The randomized controlled study will be conducted at the Ankara Yıldırım Beyazıt University Faculty of Dentistry, Department of Endodontics, and will include adult volunteers who have been diagnosed with asymptomatic apical periodontitis, present periapical lesions with PAI scores of 2, 3, and 4, have an indication for root canal treatment, meet the inclusion criteria of the study, and have provided written informed consent.

Volunteers will be randomly selected from patients attending our clinic according to lesion size. A computer-assisted randomization method (www.randomizer.org) will be used. Root canal treatments will be completed using AH Plus or TotalFill BC root canal sealers.

The required sample size will consist of a total of 64 volunteers: 16 volunteers with PAI 2-3 scored teeth treated with AH Plus, 16 volunteers with PAI 4 scored teeth treated with AH Plus, 16 volunteers with PAI 2-3 scored teeth treated with TotalFill BC, and 16 volunteers with PAI 4 scored teeth treated with TotalFill BC.

After completion of the root canal treatments, postoperative radiographs will be obtained and follow-up will be performed at 6 months. Postoperative pain will be assessed at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as at 1 week following completion of the root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged between 18 and 60 years with no systemic diseases
2. Teeth with periapical lesions (apical periodontitis) that have not undergone previous root canal treatment
3. Single-rooted maxillary and mandibular teeth
4. Teeth with PAI scores of 2, 3, and 4 according to the PAI classification
5. Teeth without a sinus tract or acute apical abscess
6. Patients who voluntarily agree to participate in the study and attend follow-up visits
7. Teeth with sufficient remaining tooth structure to allow restoration with a direct restoration after root canal treatment -

Exclusion Criteria:

Patients who have used antibiotics, analgesics, or anti-inflammatory drugs within the last 7 days

Pregnant or breastfeeding patients

Patients with traumatic malocclusion

Patients without occlusal contact

Teeth with root resorption, open apices, or calcification

Teeth presenting gingival recession greater than 3 mm, deep periodontal pockets, or mobility

Teeth with root fractures or cracks

Presence of an adjacent tooth requiring endodontic treatment that may cause referred pain

Multirooted teeth

Teeth with a PAI score of 5

Teeth requiring restorations such as endocrowns, onlays, overlays, or full crowns due to excessive loss of tooth structure after root canal treatment

Teeth with structural loss severe enough to require post-core application

Cases in which adequate anesthesia cannot be achieved with local anesthesia alone (requiring additional intrapulpal or intraligamentary anesthesia)

Teeth requiring active periodontal treatment

Individuals with severe systemic diseases

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Fractal analysis | 6. month
  In this study, fractal analysis of each sample will be performed using the box-counting method.
VAS scala | 6.,12.,24.,36.,48.,72. hours and 1 week
  Volunteers will be asked to record the pain they experience before treatment and at the 6th, 12th, 24th, 36th, 48th, and 72nd hours, as well as 1 week after treatment, on a form using the Visual Analog Scale (VAS). One week after treatment, volunteers will be contacted by telephone, and the pain scores indicated on the pain assessment forms will be obtained and recorded in the patient files.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Büşra KESKİN KESKİN, Principal Investigator — Ankara Yıldırım Beyazıt University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegde VR, Hegde SR, Fanibunda UE, Vartak MA. Comparative evaluation of postoperative pain and healing following root canal obturation with calcium silicate and bioactive glass-based sealers to epoxy resin-based sealers: A systematic review and meta-analysis. J Conserv Dent Endod. 2025 Mar;28(3):211-221. doi: 10.4103/JCDE.JCDE_8_25. Epub 2025 Mar 3. PMID 40256693
- [Background] Gotler M, Bar-Gil B, Ashkenazi M. Postoperative pain after root canal treatment: a prospective cohort study. Int J Dent. 2012;2012:310467. doi: 10.1155/2012/310467. Epub 2012 Mar 15. PMID 22505897
- [Background] de Oliveira CB, Rocha TG, Pintor AVB, Magno MB, Abrahao AC, Maia LC, Romanach MJ, Visconti MA. Using fractal analysis to assess periapical bone formation after endodontic treatment: A systematic review and meta-analysis. Imaging Sci Dent. 2025 Jun;55(2):126-138. doi: 10.5624/isd.20240221. Epub 2025 Apr 10. PMID 40607066
- [Background] Cosar M, Kandemir Demirci G, Caliskan MK. The effect of two different root canal sealers on treatment outcome and post-obturation pain in single-visit root canal treatment: A prospective randomized clinical trial. Int Endod J. 2023 Mar;56(3):318-330. doi: 10.1111/iej.13870. Epub 2022 Nov 22. PMID 36385378
- [Background] Tan HSG, Lim KC, Lui JN, Lai WMC, Yu VSH. Postobturation Pain Associated with Tricalcium Silicate and Resin-based Sealer Techniques: A Randomized Clinical Trial. J Endod. 2021 Feb;47(2):169-177. doi: 10.1016/j.joen.2020.10.013. Epub 2020 Oct 22. PMID 33098889